CLINICAL TRIAL: NCT06657677
Title: Assessing the Immediate Increase in Serum Ferritin After Oral Iron Doses: an Experimental Study in Iron-deficient Women.
Brief Title: Assessing the Immediate Increase in Serum Ferritin After Oral Iron Doses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Rigutto (Other)
Responsible Party: Sponsor-Investigator, Jessica Rigutto, PhD, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INFER Study 1
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-10

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: oral iron supplementation; serum ferritin
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 40 mg (Experimental): single dose of 40 mg oral iron
  Interventions: Dietary Supplement: 40mg oral iron dosing
- 100 mg (Experimental): single dose of 100 mg oral iron
  Interventions: Dietary Supplement: 100mg oral iron dosing
- 180 mg (Experimental): single dose of 180 mg oral iron
  Interventions: Dietary Supplement: 180mg oral iron dosing

INTERVENTIONS:
Dietary Supplement: 40mg oral iron dosing — Participants will receive a single morning oral dose of iron as Fe57-labelled ferrous sulfate
  Arms: 40 mg
Dietary Supplement: 100mg oral iron dosing — Participants will receive a single morning oral dose of iron as Fe57-labelled ferrous sulfate
  Arms: 100 mg
Dietary Supplement: 180mg oral iron dosing — Participants will receive a single morning oral dose of iron as Fe57-labelled ferrous sulfate
  Arms: 180 mg

SUMMARY:
Serum ferritin is a key indicator of body iron stores and is widely used in monitoring iron status. However, oral iron doses can acutely elevate SF levels, potentially biasing assessments of iron stores during supplementation. This study aims to investigate the extent and duration of the acute iron-induced effect on serum ferritin, as well as its protein characteristics, following the administration of a single iron dose

ELIGIBILITY:
Inclusion Criteria:

* Low iron stores (SF levels < 30 µg/L),
* no anemia (Hb > 120 g/L)
* no inflammation (CRP < 5 mg/L)
* 18 to 45 years old.
* Body weight <70 kg
* Normal body Mass Index (18.5-26.5 kg/m2)

Exclusion Criteria:

* Any chronic or acute disease
* Consumption of mineral and vitamin supplements since screening and over the study period
* Blood transfusion, blood donation or significant blood loss over the past 6 months,
* Pregnant or breastfeeding,
* Continuous/long-term use of medication during the whole studies (except for contraceptives)
* Therapeutic iron infusion over the past 6 months,
* Known hypersensitivity or allergy to iron supplements,
* Intention to become pregnant over the course of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Serum ferritin | study day 1
  Serum ferritin concentration
Serum ferritin | study day 7
  Serum ferritin concentration

SECONDARY OUTCOMES:
C-reactive protein | study day 0
  C-reactive protein concentration in serum
Serum ferritin | study day 0
  Serum ferritin concentration
Serum ferritin | study day 6
  Serum ferritin concentration
Serum ferritin | study day 14
  Serum ferritin concentration
Serum ferritin | study day 5
  Serum ferritin concentration
Serum ferritin | study day 4
  Serum ferritin concentration
Serum ferritin | study day 3
  Serum ferritin concentration
Serum ferritin | study day 2
  Serum ferritin concentration
alpha(1)-acid-glycoprotein | study day 0
  alpha(1)-acid-glycoprotein concentration in serum
soluble transferrin receptor | study day 0
  soluble transferrin receptor in serum
Hemoglobin | study day 0
  Hemoglobin concentration
Serum iron | study day 0
  serum iron concentration in circulation
Serum iron | study day 1
  serum iron concentration in circulation
Serum iron | study day 2
  serum iron concentration in circulation
Serum iron | study day 3
  serum iron concentration in circulation
Serum iron | study day 4
  serum iron concentration in circulation
Serum iron | study day 5
  serum iron concentration in circulation
Serum iron | study day 6
  serum iron concentration in circulation
Serum iron | study day 7
  serum iron concentration in circulation
Serum iron | study day 14
  serum iron concentration in circulation
Isotopic composition of Serum Ferritin | study day 0
  shift in stable iron isotopes in serum ferritin
Isotopic composition of Serum Ferritin | study day 2
  shift in stable iron isotopes in serum ferritin
Isotopic composition of Serum Ferritin | study day 7
  shift in stable iron isotopes in serum ferritin
Structural characteristics of Serum Ferritin | study day 0
  Proteomics
Structural characteristics of Serum Ferritin | study day 2
  Proteomics
Structural characteristics of Serum Ferritin | study day 7
  Proteomics
Fractional iron absorption | study day 14
  Erythrocyte iron incorporation of stable iron isotope

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stoffel, PhD, Principal Investigator — ETH Zurich
Locations (2):
- Switzerland (2):
  - ETH Zurich, Zurich, Canton of Zurich
  - Laboratory of Nutrition and Metabolic Epigenetics, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No